CLINICAL TRIAL: NCT04848103
Title: Effect of Extracorporeal Shock Wave Therapy After Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Hyun-Joong Kim, Principal investigator, Sahmyook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-1040781-A-N-012021035HR
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Rotator Cuff Injuries; Pain, Postoperative; Tissue Adhesion
MeSH Terms: conditions — Rotator Cuff Injuries; Pain, Postoperative; Tissue Adhesions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radial extracorporeal shockwave therapy (Experimental)
  Interventions: Behavioral: Radial extracorporeal shockwave therapy

INTERVENTIONS:
Behavioral: Radial extracorporeal shockwave therapy — Radial extracorporeal shockwave therapy group include Therapeutic modality(Transcutaneous electrical nerve stimulation [TENS], Microwave thermotherapy, and Superficial heat therapy), Range of motion exercise(Continuous passive motion and Active range of motion exercise).

SUMMARY:
Although radial extracorporeal shock wave therapy (rESWT) has proven to be an effective treatment, the effectiveness of the treatment has so far been controversial. There are no studies using rESWT in rehabilitation after arthroscopic rotator cuff repair (ARCR). Therefore, in this study, there is evidence that rESWT promotes pain control and healing recovery, and through previous studies, we would like to investigate whether treatment with rESWT during the intensive rehabilitation period of patients after ARCR is more effective in controlling pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old
* In case of 6 weeks after receiving arthroscopic rotator cuff repair
* When the participants wishes to enroll in the study

Exclusion Criteria:

* 65 years old or older
* If the tear area is large and augmentation is performed
* If there is a previous surgical history at the surgical site
* Osteoarthritis in the shoulder joint

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
. Pain intensity | Change from baseline pain intensity at 2 weeks
  A numeric pain rating scale (NPRS) consisting of 11 points in total from 0 points (no pain) to 10 points (the most severe pain imaginable) is used. The lower the score, the less the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Joong Kim, MSc, Principal Investigator — Principal Investigator
Locations (1):
- The Better Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HJ, Choi W, Jung J, Park S, Joo Y, Lee S, Lee S. Efficacy of radial extracorporeal shockwave therapy in rehabilitation following arthroscopic rotator cuff repair: A STROBE compliant study. Medicine (Baltimore). 2022 Sep 2;101(35):e30053. doi: 10.1097/MD.0000000000030053. PMID 36107497